

## TRIAL STATISTICAL ANALYSIS PLAN

c23146709-03

**BI Trial No.:** 1336-0011

Title: An open label phase Ib dose finding study of BI 836880 in

combination with ezabenlimab to characterize safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy in patients with locally advanced or metastatic non-squamous Non-Small

Cell Lung Cancer and in other solid tumors

Including Protocol Amendment 8 [c16151514-11]

Investigational

BI 836880

**Product(s):** Ezabenlimab (BI 754091)

Responsible trial statistician(s):

Phone:

Date of statistical

6 Jun 2022

Fax:

analysis plan:

Version: 3.0


**Proprietary confidential information** 

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

## 1. TABLE OF CONTENTS

| TITLE | PAGE1 |
|----------------|---------------------------------------------------|
| 1. | TABLE OF CONTENTS2 |
| LIST O | F TABLES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION7 |
| <b>5.</b> | ENDPOINT(S)9 |
| 5.1 | PRIMARY ENDPOINT(S) 9 |
| 5.2 | SECONDARY ENDPOINT(S)9 |
| 5.2.1 | Key secondary endpoint(s) 9 |
| 5.2.2 | Secondary endpoint(s)9 |
| 6. | GENERAL ANALYSIS DEFINITIONS13 |
| 6.1 | TREATMENT(S) |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS |
| 6.3 | SUBJECT SETS ANALYSED14 |
| | POOLING OF CENTRES |
| 6.5 | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS14 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS15 |
| 7. | PLANNED ANALYSIS |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS 16 |
| <b>7.2</b> | CONCOMITANT DISEASES AND MEDICATION16 |
| 7.3 | TREATMENT COMPLIANCE16 |
| 7.4 | PRIMARY ENDPOINT(S)17 |
| 7.5 | SECONDARY ENDPOINT(S) |
| 7.5.1 | Key secondary endpoint(s)17 |
| 7.5.2 | (Other) Secondary endpoint(s) |
| 7.7 | EXTENT OF EXPOSURE 21 |
| 7.7<br>7.8 | SAFETY ANALYSIS |
| 7.8.1 | Adverse events 22 |
| 7.8.1<br>7.8.2 | Laboratory data25 |
| 7.8.2<br>7.8.3 | Vital signs 25 |
| 7.8.3<br>7.8.4 | ECG |
| 7.0.4 | 25 |
| <u> </u> | REFERENCES |

# Boehringer Ingelheim TSAP for BL Trial No. 1336 0011

c23146709-03 

TSAP for BI Trial No: 1336-0011 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 10 | HISTORY TABLE | 32 |
|-----|----------------|------------|
| 10. | IIISTORT TADLE | J <i>L</i> |

## LIST OF TABLES

| Table 6.1: 1 | Definition of treatment periods | 13 |
|---|---|---|
| Table 7.8.1: 1 | Definitions of SSCs | 23 |
| Table 7.8.1: 2 | Definitions of SSCs from combination studies with ezabenlimab (BI | |
| | 754091) | 24 |
| | History table | |

## 2. LIST OF ABBREVIATIONS

| Term | Definition / Description |
|--------|------------------------------------------------------------|
| AE | Adverse Event |
| BHM | Bayesian Hierarchical Model |
| BOR | Best Overall Response |
| CR | Complete Response |
| CTC | Common Terminology Criteria |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DM&SM | Boehringer Ingelheim Data Management And Statistics Manual |
| DLT | Dose Limiting Toxicity |
| DoR | Duration of Response |
| DRA | Drug Regulatory Affairs |
| DMG | Dictionary Maintenance Group |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EMEA | European Agency For The Evaluation Of Medicinal Products |
| FAS | Full Analysis Set |
| GBM | Glioblastoma |
| GEP | Gene-Expression Profile |
| ICH | International Conference On Harmonisation |
| IPD | Important Protocol Deviation |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary For Regulatory Activities |
| MQRM | Medical Quality Review Meeting |
| NOA | Not Analysed |
| NOR | No Valid Result |
| NOS | No Sample |
| NSCLC | Non-Small Cell Lung Cancer |
| OR | Objective Response |

| 1 3 | |
|--------|-----------------------------------------------|
| Term | Definition / Description |
| OS | Overall Survival |
| PD | Protocol Deviation |
| PFS | Progression-Free Survival |
| PFS6 | Six-Month Progression-Free Survival |
| PK | Pharmacokinetics |
| PKS | PK Analysis Set |
| PPS | Per Protocol Set |
| PR | Partial Response |
| PSTAT | Project Statistician |
| PT | Preferred Term |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| RANO | Response Assessment in Neuro-Oncology |
| RECIST | Response Evaluation Criteria In Solid Tumours |
| REP | Residual Effect Period |
| RP2D | Recommended Phase 2 Dose |
| RPM | Report Planning Meeting |
| SA | Statistical Analysis |
| SD | Standard Deviation |
| SMC | Safety Monitoring Committee |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| SSC | Special Search Category |
| TCM | Trial Clinical Monitor |
| TESS | Treatment Emergent Signs And Symptoms |
| ToC | Table of Contents |
| TMW | Trial Medical Writer |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |

## 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, and randomization.

SAS® Version 9.4 or the latest version will be used for analyses.

R Version 3.5.1 and JAGS Version 4.3.0 or the latest versions will be used for the BLRM and BHM analyses.



## 5. ENDPOINT(S)

This is a Phase Ib study containing two parts: Part 1 (dose escalation of BI 836880 in combination with ezabenlimab (BI 754091)) and Part 2 (expansion at the RP2D in 8 cohorts with different tumour types and line of therapy) in patients with locally advanced or metastatic non-squamous NSCLC and in other solid tumors.

The primary objective for Part 1 is to determine the safety and tolerability of BI 836880 in combination with ezabenlimab and find the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D).

The primary objective for Part 2 is to assess the anti-tumor activity of BI 836880 in combination with ezabenlimab in patients with locally advanced or metastatic non-squamous NSCLC and in other solid tumors.

## 5.1 PRIMARY ENDPOINT(S)

#### PART 1:

The primary endpoint is the number of patients with dose limiting toxicities (DLTs) within the MTD evaluation period, which will be assessed for dose escalation in order to determine the maximum tolerated dose (MTD) of the combination of BI 836880 and ezabenlimab.

The MTD is defined as the highest dose with less than 25% risk of the true DLT probability being above 33% and may be considered reached if the probability that the true DLT rate is in the target interval (16%-33%) is sufficiently large during the MTD evaluation period.

The definition of DLTs for solid tumour patients is provided in Section 5.2.6.1 of the CTP.

The MTD evaluation period is defined as the time from the first administration of study treatment to the start of the second treatment cycle, i.e., the first treatment cycle.

#### **PART 2:**

The primary endpoint is Objective Response (OR) defined as best overall response (RECIST 1.1) of complete response (CR) or partial response (PR) from first treatment infusion until the earliest of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent. In the case of recurrent glioblastoma (GBM), tumour assessment will be based on RANO (Response Assessment in Neuro-Oncology) criteria.

## 5.2 SECONDARY ENDPOINT(S)

## 5.2.1 Key secondary endpoint(s)

This section is not applicable, as no key secondary endpoint has been specified in the protocol.

## 5.2.2 Secondary endpoint(s)

## **PART 1:**

- Adverse events (AEs), drug related AEs, drug related AEs leading to discontinuation during treatment period.
- Pharmacokinetic parameters C<sub>max</sub>, T<sub>max</sub>, and AUC<sub>0-504h</sub> after the first and fourth infusion cycle.

#### **PART 2:**

- Adverse events (AEs), drug related AEs, drug related AEs leading to discontinuation during treatment period.
- Disease control (DC), defined as best overall response of CR, PR, or stable disease (SD) by RECIST 1.1 (RANO for the GBM cohort) from start of treatment infusion until the earliest of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, lost to follow-up, or withdrawal of consent.
- Duration of objective response (DoR), defined as the time from first documented CR or PR by RECIST 1.1 (RANO for the GBM cohort) until the earliest of disease progression or death among patients with OR.
- Progression-free survival (PFS) (RANO for the GBM cohort and RECIST 1.1 for all other cohorts), defined as the time from first treatment infusion until disease progression or death from any cause, whichever occurs earlier.
- Tumor shrinkage (in millimeters), defined as the difference between the minimum post-baseline sum of diameters of target lesions (longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of diameters of the same set of target lesions. In GBM, using RANO criteria, tumor shrinkage will be calculated based on the difference between the post-baseline and baseline measurements of the sum of product of the largest bi-dimensional measurements for all target lesions.
- Pharmacokinetic parameters C<sub>max</sub>, T<sub>max</sub>, and AUC<sub>0-504h</sub> after the first infusion cycle.





## 6. GENERAL ANALYSIS DEFINITIONS

## 6.1 TREATMENT(S)

In this open-label Phase Ib trial, treatments are not randomized. In the dose escalation part (Part 1), the starting dose combination is BI 836880 360 mg + ezabenlimab (BI 754091) 240 mg every three weeks. Dose escalation is only performed for BI 836880. Ezabenlimab is fixed at dose 240 mg. Dose escalation decisions will be made by the Safety Monitoring Committee (SMC). Based on the dose escalation data in Part 1, the SMC will select one combination dose for the expansion cohorts in Part 2. Data of the dose expansion part (Part 2) will be displayed separately for each of the multiple cohorts.

For the dose escalation part (Part 1), the initial trial medication (i.e., dose level) assigned at the beginning of the first treatment cycle will be used as the label of the analysing treatment.

For safety analyses, adverse events (AEs) will be displayed separately within the following time periods: "Screening", "On-treatment", or "Post-study" (see Table 6.1: 1). This will be applied for both AEs and immune-related AEs. Refer to CTP Section 5.2.7.2 for details of AE collection and reporting.

Table 6.1: 1 Definition of treatment periods

| Analysing Treatment<br>Period | Start Date (including) | Stop Date (excluding) |
|---|---|---|
| Screening | Date of informed consent | The date of first trial medication administration - 1 day |
| On-treatment | Date of first administration of trial medication | Date of last trial medication<br>administration + REP, or<br>death, or DBL date,<br>whichever comes first<br>i.e., actual on-treatment<br>period + REP, |
| Post-study | Last day of on-treatment period +1 day | Date of the last contact date or death, or DBL date, whichever comes first |

Note: A 42-day residual effect period (REP) is defined for both Parts 1 and 2.

## 6.2 IMPORTANT PROTOCOL DEVIATIONS

A protocol deviation (PD) is important if it affects the rights or safety of the study patients, or if it can potentially influence the primary outcome measurements in a non-negligible way. Important protocol deviations (IPDs) are stored in the DV domain template (Excel spreadsheet). IPDs will be reviewed at Medical Quality Review Meetings (MQRMs) conducted periodically during the trial. A list of PDs will be discussed at the report planning meetings (RPMs).

If the data show other IPDs, this table will be supplemented accordingly at MQRMs or RPMs or through team review of the manual PD log. The final list of IPDs will be confirmed at the

last RPM before DBL. The decision whether a patient will be excluded from the analysis will be made at the final RPM prior to DBL.

Patients with an IPD will be identified and reported in the CTR. In addition, a per protocol set excluding patients with IPDs that could potentially impact the evaluation of the primary endpoint(s) may be defined. Primary endpoint analysis may be performed based on the per protocol set in addition to the treated set.

#### 6.3 SUBJECT SETS ANALYSED

## **Screened Set (SCS)**

This patient set includes all patients who have signed the informed consent. The screened set will be used for patient disposition tables.

## Treated set (TS)

This patient set includes all patients enrolled in the trial who were documented to have received at least one dose of ezabenlimab or BI 836880. The TS is used for both efficacy analysis and safety analyses.

## MTD set

This patient set includes all patients enrolled in dose escalation and confirmation of MTD cohort of the trial (Part 1) who were documented to have received at least one dose of ezabenlimab or BI 836880and were evaluable for the MTD determination.

## **Expansion cohort treated set**

This patient set includes all patients enrolled in the expansion part (Part 2) and were documented to have received at least one dose of ezabenlimab or BI 836880.

## PK analysis set (PKS)

This patient set includes all patients in the TS who provide at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviation. PKS is used for statistical PK analysis.



## 6.5 POOLING OF CENTRES

This section is not applicable because centre is not included in the statistical model.

## 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates") (3). Missing data and outliers of PK data are handled according to (2). Please refer to Section 7.5 of the CTP for more details. According to (2), missing biomarker data (NOS - no sample, NOR - no valid result, NOA - not analyzed) will not be imputed. Handling of data below or above the limit of quantification, e.g., the myriad panel data:

• BLQ data will be replaced by ½ LLOQ.

• ALQ data will be replaced by ULOQ, if ULOQs are available. Otherwise, ALQ data will be excluded from the analysis.

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

#### Visit labels

Study days and visits will be labelled according to the flow charts in the CTP. The visit schedule with accompanying details can also be found in the flow charts in the CTP.

## **Definition of "baseline"**

For laboratory values, the baseline value is the <u>most recently observed value before or on the first day of infusion of trial medication</u>; for laboratory measurements, the examination time may also need to be considered, in instances where time is recorded in addition to date. For all other data values, baseline is defined as <u>the most recent measurement taken prior to first administration of trial medication</u>. If not available, then the values reported at the screening visit will be considered.

#### Time windows

Time windows and visits will be calculated to determine the planned day of tumour measurement and response status based on the protocol-specified tumour imaging schedule. Imaging data will be displayed as: Screening, Week 6, Week 12, Week 18, etc. The number of weeks will be calculated using their relative day (from start of treatment) using a ±3 week window. (Images taken in the first 3 weeks from start of treatment will be assigned to Week 6.) Images which are not older than 28 days at start of treatment will be sufficient as screening images and do not need to be repeated.

#### How to include measurements taken between time windows

The same visit windows will be used for safety laboratory and vital sign assessments. If there are multiple safety or laboratory values in one time window on treatment, the worst value will be selected for the by-visit analyses.

## 7. PLANNED ANALYSIS

For End-Of-Text (EoT) tables, the set of summary statistics includes: N / Mean / SD / Min / Q1 (lower quartile) / Median / Q3 (upper quartile) / Max.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not).

Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

## 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.

## 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report.

Compliance will be calculated for subjects having attended the visit. A subject is considered having attended the visit if the indicated visit is captured in the eCRF database. In particular, if a subject attended the visit, but is not treated at the visit, the compliance of this visit is considered as 0%.

Compliance with trial medication will be based on the drug infusion/administered eCRF data and calculated as amount of drug infused/administered divided by the amount of drug to be infused/administered expressed as a percentage, see calculations below.

"Per Visit" compliance to trial medication will be calculated as follows:

 $\frac{\text{(Amount of drug infused/administered at Visit X(n))}}{\text{(Amount of drug planned to be infused/administered at Visit X(n))}} \times 100$ 

Overall compliance for first treatment cycle of all patients will be calculated as mean of "per visit" compliance at visit Day 1.

Overall compliance for second treatment cycle onwards (from Day 22 onwards) of all patients will be calculated as mean of "per visit" compliance at each visit. Overall compliance to trial medication will be calculated as mean of the "per visit" compliance.

The compliance will be based on the total volume infused in mL (eCRF data) compared to total volume prepared (eCRF data).

## 7.4 PRIMARY ENDPOINT(S)

The analysis of primary endpoints will be performed as defined in the CTP with the approach proposed by Berry et al. (2013). Posterior distributions for the ORRs will be summarized with Mean, Median, 2.5%, and 97.5 % quantiles.

## 7.5 SECONDARY ENDPOINT(S)

The analysis of secondary endpoints will be performed as defined in the CTP.

## 7.5.1 Key secondary endpoint(s)

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 (Other) Secondary endpoint(s)

Not applicable.



#### 7.7 **EXTENT OF EXPOSURE**

Treatment exposure will be primarily summarized by the total on-treatment time and has been defined in Section 5.4 of this TSAP.

Treatment interruptions before permanent discontinuation will not be excluded. In Part 1, summary statistics for treatment time by each dose level and the dosage of BI 836880 over time will also be provided.

## 7.8 SAFETY ANALYSIS

The safety analyses will be performed as defined in the CTP. All safety analyses will be performed on the treated set of Part 1 and Part 2 of this trial.

## 7.8.1 Adverse events

The analyses of adverse events (AE) will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and not on the number of AEs. Two analyses will be performed. The first analysis of safety will be performed for the first part of the trial (determination of the MTD/RP2D, first cycle only, dose level = initial dose at the start of the treatment, treated set). This descriptive analysis will evaluate the MTD/RP2D. The second analysis will be performed with respect to all cycles for part 1 and will act as a support for the determination of the MTD/RP2D (treated set).

For analysis of duration, severity, etc. of multiple AE occurrences, data on the case report form (CRF) will be collapsed into AE episodes provided that all of the following applies:

- The same MedDRA lowest level term was reported for the occurrences.
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence).
- Treatment did not change between the onset of the occurrences or treatment changed between the onsets of the occurrences, but no deterioration was observed for the later occurrence.

For further details on summarization of AE data, please refer to the guideline 'Handling and summarization of adverse event data for clinical trial reports and integrated summaries' (5).

For patients treated with the test drug, that means that all adverse events occurring between first drug infusion and the REP after last drug infusion or death, whichever occurs first, will be assigned to the on-treatment period. All adverse events occurring before any study drug infusion will be assigned to 'screening' and all adverse events occurring after last study drug infusion + the REP will be assigned to 'post-study' (for listings only). For details on the treatment definition, see Section 6.1.

An overall summary of adverse events will be presented. This summary will exclude the rows 'Severe AEs', 'Significant AEs' and 'Other significant AEs' but will include additional rows for 'AEs leading to dose reduction', 'AEs leading to death' and 'AEs by highest Common Terminology Criteria (CTC) grade'.

Additional AE tables will be produced for AEs of special interest (hepatic injury as defined in CTP Section 5.2.7.1 and DLTs as defined in CTP Section 5.2.6.1), providing further details on highest CTC grade, action taken with study drug, and time to first onset of AE.

The frequency of patients with adverse events will be summarized by maximum CTC grade (grades 1, 2, 3, 4, 5 and all grades), treatment, primary system organ class and preferred term for each of the following AE tables as well as relatedness of AEs to treatment and seriousness:

• All AEs

- Drug-related AEs
- Immune-related AEs
- AEs leading to dose reduction
- Drug-related AE leading to dose reduction
- Immune-related AEs leading to dose reduction
- AEs leading to treatment discontinuation
- Drug-related AEs leading to treatment discontinuation
- Immune-related AEs leading to treatment discontinuation
- Drug-related AEs leading to treatment discontinuation or dose reduction
- Immune-related AEs leading to treatment discontinuation or dose reduction
- AEs leading to death
- Serious AEs
- Drug-related serious AEs
- AESIs
- DLTs (in Part 1 dose escalation only)

All tables will be sorted by system organ class (SOC) according to the standard sort order specified by the European Medicines Agency (EMA). Preferred terms (PTs) will be sorted by frequency (within SOC).

The above tables will be repeated with the project-defined grouping of AE terms. Details of the project-defined groupings are defined in the technical TSAP. In these tables, the grouped AEs will replace the original PTs for all AEs that are included within the grouped term. The grouped AE categories will then be tabulated along with all remaining MedDRA PTs, sorted by descending frequency.

A reference table presenting the entire project defined groupings and MedDRA PTs within each grouping will also be produced.

The frequency of patients with user defined AEs will be presented by special search category, preferred term, and highest CTCAE grade. Special search categories (SSCs) for AEs are defined in Table 7.8.1: 1 below.

Table 7.8.1: 1 Definitions of SSCs

| N | Medical concept | Definition (for programmers) | Other monitoring options |
|---|---|---|---|
| 1 | Fatigue / asthenia | HLT 10003550 | |
| 2 | Hypertension | SMQ 20000147 | Narrow |
| 3 | Proteinuria | SMQ 20000220 | Narrow |
| 4 | Haemorrhage | SMQ 20000040 | Narrow |
| | | SMQ 20000039 | Narrow |
| 5 | Embolic and thrombotic events | SMQ 20000081 | Narrow |
| | | SMQ 20000115 | Narrow and broad |
| 6 | GI perforation | SMQ 20000107 | Narrow |

| N | Medical concept | Definition (for programmers) | Other monitoring options |
|---|---|---|---|
| 7 | Infusion related reactions | SMQ 20000021 | Narrow |
| | | + PT 10051792 | |
| | | + PT 10082742 | |
| 8 | Cardiac failure | SMQ 20000004 | Narrow and broad |

Additional SSCs for AEs that are to be completed for combination studies with ezabenlimab (BI 754091) are defined in Table 7.8.1: 2 below.

Table 7.8.1: 2 Definitions of SSCs from combination studies with ezabenlimab (BI 754091)

| N | Term | Definition# | SMQ code |
|---|---|---|---|
| 1 | Non-infectious diarrhoea | Noninfectious diarrhea (SMQ) Broad | 20000218 |
| 2 | Drug related hepatic disorders | Drug related hepatic disorders -<br>comprehensive search (SMQ) Broad | 20000005 |
| 3 | ILD | Interstitial lung disease (SMQ) Narrow | 20000042 |
| 4 | Thyroid dysfunction | Thyroid dysfunction (SMQ) Broad | 20000159 |
| 5 | SCAR | Severe cutaneous adverse reactions (SMQ) Broad | 20000020 |
| 6 | Peripheral neuropathy | Peripheral neuropathy (SMQ) Broad | 20000034 |
| 7 | Non-infectious meningitis | Noninfectious meningitis (SMQ)<br>Broad | 20000134 |
| 8 | Non-infectious encephalitis | Noninfectious encephalitis (SMQ)<br>Broad | 20000132 |
| 9 | Acute renal failure | Acute renal failure (SMQ) Broad | 20000003 |
| 10 | Cardiomyopathy | Cardiomyopathy (SMQ) Broad | 20000150 |
| 11 | Guillain-Barre syndrome | Guillain-Barre syndrome (SMQ) Broad | 20000131 |
| 12 | Haematopoietic cytopenias | Haematopoietic cytopenias (SMQ)<br>Broad | 20000027 |
| 13 | Acute pancreatitis | Acute pancreatitis (SMQ) Broad | 20000022 |
| 14 | Cardiac arrhythmias | Cardiac arrhythmias (SMQ) Broad | 20000049 |
| 15 | Heart failure | Cardiac failure (SMQ) Narrow | 20000004 |
| 16 | Vasculitis | Vasculitis (SMQ) Narrow | 20000174 |

<sup>#</sup> This column indicates whether the Term(s) provided in the first column are MedDRA preferred terms (PT), Standardised MedDRA Queries (SMQ), or BI customized MedDRA Queries (BIcMQ).

## 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (7). CTC grade for applicable lab parameters will be calculated according to CTCAE v5.0 (6).

Descriptive statistics of all converted laboratory values by visit will be provided including changes from baseline. Frequency tables of transitions relative to the reference range and of possible clinically significant abnormalities will be produced. For those parameters that have CTC grading possible clinically significant abnormalities are defined as those laboratory values with a CTC grade  $\geq 2$  that have had an increase of  $\geq 1$  grade from baseline. For those parameters for which no CTC grade has been defined standard BI project definitions will be used to decide on clinical significance. Further frequency table will show the transition of CTC grade from baseline to worst value and from baseline to last value on treatment.

Summaries will be produced of laboratory data recorded prior to treatment, on-treatment and post-treatment. For details on the treatment definition, see Section 6.1.

The focus of the laboratory data analysis will be on the following laboratory parameters:

- Low values: Activated Partial Thromboplastin Time (aPTT), Prothrombin Time (PT), International Normalised Ratio (INR), White Blood Cell Count (WBC) with differential, Platelets (PLT)
- High values: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), bilirubin, Alkaline Phosphatase (AP), Activated Partial Thromboplastin Time (aPTT), Prothrombin Time (PT), International Normalised Ratio (INR), Protein levels in urine

## 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report. A shift table will be provided for change from baseline over the course of treatment for systolic and diastolic blood pressure.

## **7.8.4** ECG

ECG data will be collected as described in CTP Section 5.2.4. Clinically significant findings in ECG data will be reported under "Adverse events" if applicable and will be analysed accordingly. In addition, patients with abnormal overall assessments at any time on treatment will be summarized in a descriptive manner.





#### 8. **REFERENCES**

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic |
|---|---|
| | E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
| 2 | 001-MCS 36-472: "Standards and processes for analyses performed within Clinical |
| | Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 3 | 001-MCG-156_RD-01: "Handling of missing and incomplete AE dates", current |
| | version; IDEA for CON. |
| 4 | 001-MCG-420: "Statistical Methods for Pharmacokinetics", Version 3.0, IDEA for |
| | CON. |
| 5 | 001-MCG-156: "Handling and summarization of adverse event data for clinical trial |
| | reports and integrated summaries", current version; IDEA for CON. |
| 6 | Common Terminology Criteria for Adverse Events (CTCAE): version 5.0, published: |
| | November 27, 2017 (v5.0) |
| | https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5 |
| | _Quick_Reference_5x7.pdf (access date: April 14, 2020), U.S. Department of Health |
| | and Human Services, National Institutes of Health, National Cancer Institute 2017. |
| 7 | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current |
| | version; IDEA for CON. |

## 10. HISTORY TABLE

Table 10: 1 History table

This is a revised TSAP including the following modifications.

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial | 18-APR-2018 | | None | This is the initial TSAP with necessary information for trial conduct. |
| Revised | 17-APR-2020 | | Sections 2, 5, 6, 7, 8 | This is a revised TSAP with revisions reflecting changes in CTP version 5.0. |
| Revised | 26-OCT-2020 | | | |
| Revised | 19-MAR-2021 | | | |

| | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Revised | 23-AUG-2021 | | | |
| Revised | 05 MAN 2022 | | | |
| Revised | 05-MAY-2022 | | | |
| | | _ | | |
| Final | DD-MMM-YY | XX | XX | This is the final TSAP. |



## APPROVAL / SIGNATURE PAGE

Document Number: c23146709 Technical Version Number: 3.0

**Document Name:** 8-01-tsap

**Title:** An open label phase Ib dose finding study of BI 836880 in combination with ezabenlimab to characterize safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy in patients with locally advanced or metastatic non-squamous Non-Small Cell Lung Cancer and in other solid tumors

## **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval-Team Member Medicine | | 28 Jun 2022 22:30 CEST |
| Approval-Clinical Trial Leader | | 29 Jun 2022 08:21 CEST |
| Approval-Medical Writer | | 29 Jun 2022 11:42 CEST |
| Approval-Project Statistician | | 29 Jun 2022 14:33 CEST |
| Approval-Translational Medicine<br>Expert | | 30 Jun 2022 04:15 CEST |
| Approval-Clinical Pharmacokinetics | | 30 Jun 2022 16:36 CEST |

**Boehringer Ingelheim Document Number:** c23146709 **Technical Version Number:**3.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|